CLINICAL TRIAL: NCT04135378
Title: Effect of Low Doses of Vitamin C on Salivary Cortisol , Heart Rate , Blood Pressure During Group Presentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Ali A. Al-fahham, Assistance Professor, Kufa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KufaU2
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Stress, Psychological
Keywords: vitamin C , salivary cortisol , heart rate , blood pressure
MeSH Terms: conditions — Stress, Psychological | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Experimental randomized placebo trial study approach was designed to meet the previously mentioned objectives of the current study. The period of the study is from 1st November 2018 to 20th April 2019. A random sample of (90) students was taken in this study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- student- ascorbic acid (Experimental): Student that have presentation given ascorbic acid ( 500 mg per day) for one week before presentation .
  Interventions: Drug: ascorbic acid
- Control- ascorbic acid like (Placebo Comparator): ascorbic acid like placebo for one week before presentation
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ascorbic acid — Study Group :- ascorbic acid ( 500 mg per day) for one week before presentation
  Other Names: vitamin C
  Arms: student- ascorbic acid
Other: placebo — :- included 30 students given placebo for one week before presentation.
  Arms: Control- ascorbic acid like

SUMMARY:
Vitamin C (ascorbic acid) is a well-known antioxidant that is involved in anxiety, stress, depression, fatigue and mood state in humans . The purpose of this study is to investigate the effect of low doses of vitamin C on decreasing the level of public speaking stress in term of salivary cortisol , blood pressure (systolic and diastolic) and heart rate . A purposive sample of (90) were included in this randomized placeboled trial study (60 students were given 500 mg of vitamin c per day for one week a group presentation while 30 other students were given placebo for one week before a group presentation) . Salivary cortisol was measured by means of commercial immunoenzymatic kits . Blood pressure (systolic and diastolic) and heart rate were measured immediately before and after presentation .

DETAILED DESCRIPTION:
Experimental randomized placebo trial study approach was designed to meet the previously mentioned objectives of the current study. The period of the study is from 1st November 2018 to 20th April 2019. A random sample of (90) students was taken in this study .

The students were divided in to two groups :-

1. Study Group :- included 60 students given vitamin C ( 500 mg per day) for one week before presentation .
2. Placebo :- included 30 students given placebo for one week before presentation. Exclusion criteria included : chronic diseases (DM , hypertension), hormonal disturbances, psychotic disorders, kidney stones and anemia . Students that have previous experience of public speaking were also excluded .

Participants were asked to rinse their mouth with water before collecting saliva. A minimum volume of 1 mL saliva was obtained directly by expectorating into a collecting tube. Food and beverages such as tea, soft drinks, and coffee were not permitted 30 minutes prior to any sample collection. Because salivary cortisol concentration is independent of flow rate and sugarless gum does not interfere with the salivary assay, 21 participants were permitted to chew sugarless gum if needed to stimulate saliva flow. Participants were also instructed not to brush their teeth 30 minutes before saliva collection and to refrain from wearing lipstick on the day of saliva collection (Hellhammer et al., 1987) .

ELIGIBILITY:
Inclusion Criteria:

- students have a presentation

Exclusion Criteria:

- Exclusion criteria included : chronic diseases (DM , hypertension), hormonal disturbances, psychotic disorders, kidney stones and anemia . Students that have previous experience of public speaking were also excluded .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Cortisol | for six months
  levels of cortisol in saliva between 3-19 microg/l

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Al-fahham, Asst. Prof., Principal Investigator — Kufa University
Locations (1):
- Kufa University, Najaf, Kufa, Iraq

IPD SHARING:
Plan to Share IPD: No